CLINICAL TRIAL: NCT05389956
Title: Identification of Risk Factors for Cardiovascular Disease and Cancer in Korean Population: A Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Sangwoo Park, MD, Ulsan University Hospital
Other Study IDs: 2021-12-014-003
Record Dates: First submitted 2022-05-21; First posted 2022-05-25 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases; Malignancy; Risk Factor
Keywords: Cardiovascular disease; Malignancy; Risk factor
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ulsan University Hospital-Health Screening Cohort (UUH-HEALS): Ulsan University Hospital-Health Screening Cohort is a prospective cohort of participants who participated in general health screening programs at the Health Promotion Center of Ulsan University Hospital (Ulsan, South Korea). This cohort includes health screening participants aged 19 years and older from community and workplace. The purpose of this cohort is to offer relevant and useful data on health risk factors in the field of non-communicable diseases such as cardiovascular disease and malignancy.

SUMMARY:
Cancer and cardiovascular disease are the global leading causes of death. These two disease entities are multifactorial disease that are caused by several factors. The aim of this prospective cohort study was to investigate the status of risk factors profiles and health related behavior in Korean population, and to discover novel risk factors associated with the occurrence of endpoint events.

DETAILED DESCRIPTION:
This is a single center, observational, prospective cohort study. The primary outcomes include the incidence of MACE (major adverse cardiovascular events) and the incidence of any malignancy. We plan to collect the baseline information at enrollment and the occurrence of clinical endpoint events will be followed for at least 10 years. The study will enroll 510,000 subjects aged ≥19 years who underwent a general health screening in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 19 years and older who underwent a general health screening at the health promotion center of Ulsan University Hospital (Ulsan, Korea)
* Subjects have to agree to participate by signing a consent

Exclusion Criteria:

* Subjects who cannot or reject to sign the consent form.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health screening participants aged 19 years and older from community and workplace
Sampling Method: Probability Sample
Enrollment: 510000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2042-08 (Estimated); Study Completion 2052-08 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular event (MACE) | 10 year
  A major adverse cardiovascular event (MACE) of cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke
Incidence of malignancy | 10 year
  The occurrence of any malignancy of interest

SECONDARY OUTCOMES:
All-cause death | 10 year
Cardiovascular death | 10 year
Myocardial infarction | 10 year
Stroke | 10 year
Cancer related mortality | 10 year

CONTACTS AND LOCATIONS:
Overall Officials: Sangwoo Park, MD, Principal Investigator — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided